CLINICAL TRIAL: NCT07245147
Title: REDO-AF: Randomized Evaluation of Dual Options for AF Re-intervention
Acronym: REDO-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jacqueline Joza (Other)
Responsible Party: Sponsor-Investigator, Jacqueline Joza, Cardiac Electrophysiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-37-2025-11136
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF); AV Node Ablation; Left Bundle Branch Pacing
Keywords: Atrial fibrillation; pace and ablate; AV node ablation; Left bundle branch pacing; LBBP; Redo
MeSH Terms: conditions — Atrial Fibrillation | interventions — Furin

STUDY DESIGN:
Intervention Model Description: The REDO AF Trial is a prospective, randomized, controlled, open-label multicenter study design (PROBE) with 1:1 randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): LBBP + AV Node ablation
  Interventions: Procedure: Pace and Ablate
- Control (Active Comparator): Redo AF ablation
  Interventions: Procedure: Redo AF Ablation

INTERVENTIONS:
Procedure: Redo AF Ablation — Redo AF Ablation as per operator discretion
  Arms: Control
Procedure: Pace and Ablate — Left bundle branch pacing with AV node ablation
  Arms: Experimental

SUMMARY:
The goal of this randomized open-label clinical trial is to evaluate two different strategies for the treatment of recurrent atrial fibrillation (AF) after AF ablation. Patients who have symptomatic, drug-refractory recurrence of AF will be randomized to either a redo AF ablation vs conduction system pacing with AV node ablation. Patients will need to have undergone at least 1 prior AF ablation to be considered eligible for the study. The current trial is a vanguard study of 16 patients and will determine the feasibility of enrolment, compare changes in quality of life, and inform the design of the definitive REDO AF trial.

DETAILED DESCRIPTION:
Recurrence rates after atrial fibrillation (AF) ablation procedures are high at approximately 50% at 18 months and are associated with procedural risk as well as with significant costs. There is limited guidance on how best to treat those who recur post AF ablation. The combination of pacemaker implantation and atrioventricular node ablation (AVNA), so-called "pace-and-ablate" strategy, is an alternative treatment in patients who are at high risk of AF recurrence, especially since the recent introduction of left bundle branch pacing (LBBP). LBBP is a type of pacing strategy that captures the intrinsic conduction system and preserves normal physiological ventricular activation. The REDO-AF Trial will compare a strategy of pace-and-ablate therapy with LBBP + AVNA as compared to a strategy of redo AF ablation in medically refractory patients presenting with recurrent symptomatic AF post AF ablation. We hypothesize that a pace-and-ablate strategy will result in reduction in cardiovascular hospitalizations, procedural complications and an improvement in quality of life (QOL). The definitive research question of the REDO-AF trial is: Can a strategy of LBBP combined with AVNA in patients with recurrent, symptomatic, drug-refractory AF after previous AF ablation(s), who remain at high risk of recurrence, lead to a reduction in cardiovascular hospitalizations, reduction in procedure or device-related complications, and a greater improvement in QOL as compared to a subsequent (redo) AF ablation.

ELIGIBILITY:
Inclusion Criteria:

* One or more prior left atrial (LA) ablation procedure(s) for AF
* Symptomatic AF/atypical atrial flutter/atrial tachycardia with failure of or intolerance to medical rate or rhythm control therapy, that is detected at >2 months post most recent LA ablation procedure
* Either a LA volume index on any prior echo of >= 45ml/m2 or LA diameter >= 50mm OR a HATCH score >=2 (where 1 point is given for each for hypertension, Age>75, COPD, and 2 points for each of stroke/TIA, or HF (defined as signs or symptoms of pulmonary edema and may include HFrEF or HFpEF)
* Be considered suitable for both treatment strategies of redo ablation and pacemaker and AV node ablation
* Willingness to participate, complete the QOL questionnaires and ability to sign informed consent

Exclusion Criteria:

* Severe valvular disease defined by echo criteria
* Myocardial infarction, stroke, or coronary revascularization within the previous 3 months
* LVEF <40% or need for an ICD
* Life expectancy <24 months
* Lack of capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Cardiac Hospitalization | 1 year
  cardiovascular hospitalization defined as a greater or equal to 24 hour stay in hospital due to heart failure, myocardial infarction, stroke/transient ischemic attack or systemic embolism, arrhythmia recurrence, or complications related to the procedure or device implant that require hospitalization), or a hospital visit (of any duration) for re-intervention.
Quality of Life Improvements | 1 year
  MLHFQ
Feasibility of Enrolment | 1 year
  Feasibility of Enrolment
Procedural and Device-Related Complications not requiring a hospitalization | 1 year
  Component of the Definitive Trial; collected as a secondary endpoint for the vanguard

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Canada

IPD SHARING:
Plan to Share IPD: Yes